CLINICAL TRIAL: NCT03271814
Title: Brain Biomarker on Inflammation Response
Acronym: LPS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI moved to another institution before enrollment could start.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, L. Elliot Hong, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HP-00076657
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- LPS-Patient (Experimental): Schizophrenia patients who are randomized to receive LPS injection.
  Interventions: Biological: LPS
- LPS-Healthy (Active Comparator): Healthy controls who are randomized to receive LPS injection.
  Interventions: Biological: LPS
- Placebo-Patient (Placebo Comparator): Schizophrenia patients who are randomized to receive placebo injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: LPS — 0.6 by/kg LPS single dose iv
  Arms: LPS-Healthy; LPS-Patient
Other: Placebo — Sterile Water
  Arms: Placebo-Patient

SUMMARY:
In a double-blinded, randomized, parallel controlled design, patients with schizophrenia spectrum disorder will be exposed to a single dose of lipopolysaccharide (LPS) (LPS-patient). Clinical symptoms, blood samples, and brain imaging will be assessed at baseline and after LPS. There will be two comparison groups. Comparison groups include an age- and sex-matched healthy control group also exposed to the same LPS (LPS-control), and an age- and sex-matched sample of patients with schizophrenia on placebo (Placebo-patient). As in Phase I studies, multiple interim analyses are expected so the current design may be modified, which will be communicated during annual reports (21CFR312.30).

DETAILED DESCRIPTION:
Schizophrenia spectrum disorders are a major public health burden due to functional and cognitive impairment, psychosis and other symptoms, and high comorbidity. Unfortunately, current therapies have limited effectiveness in treating some of the symptoms and most of the cognitive deficits. Alternative biological models of the disease are needed for developing new and more effective treatment. Neuroinflammation has increasingly been implicated in the pathophysiology of schizophrenia. Patients with schizophrenia have signs of low-grade, chronic inflammation, including elevated blood levels of pro-inflammatory cytokines and other immune markers. Administration of LPS is the standard immune challenge to investigate the body's immune response in a wide range of disorders. Our goal is to use LPS to investigate whether schizophrenia patients have abnormal immune response to LPS and whether the abnormality is associated with specific brain imaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55
2. Patients must be on antipsychotic medication and clinically stable, defined as no hospitalization or major change in antipsychotic medication in the past 4 weeks
3. Patients must pass the ESC with score 10 or above
4. BMI 35 or less -

Exclusion Criteria:

1. History of major medical illness including, but not limited to, history of heart attack, stroke, TIA (transient ischemic attack)
2. History of organic brain disorders that may affect neurophysiological measurements, including seizure disorder, brain tumor, head injury with evidence of significant cognitive deterioration
3. DSM diagnosis of substance use disorder within 6 months except nicotine and marijuana
4. Prior suicide attempt or frequent suicidal ideations, or current suicidal ideation assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
5. Women who have positive urine pregnancy tests; Women who plan to become pregnant, or are breastfeeding
6. Frequent (more than once) history of syncope (fainting) of unknown reason
7. Unable to undergo MRI scanning due to metallic devices or objects or claustrophobia
8. Presence of co-morbid inflammatory disorders such as rheumatoid arthritis
9. Presence of acute or chronic infection; have received flu or similar vaccine in the past 4 weeks
10. Current regular use of non-steroidal anti-inflammatory drugs or immune modifying drugs
11. Clinically significant abnormalities on screening laboratory tests
12. Blood pressure <90/60 or > 150/100, or pulse <55 or > 100 beats/minute, or temperature > 99.5°F
13. 12-Lead ECG demonstrating QTcF >450 msec or a QRS interval >120 msec. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF values should be used to determine the subject's eligibility

    -

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
IL-6 | Hourly for 6 hours
  Cytokine IL-6 at baseline and response to LPS challenge (to be reported in pg/ml or IU/ml)

SECONDARY OUTCOMES:
Brain imaging structure and function via MRI | 3 to 6 hours
  Brain imaging at baseline and response to LPS challenge (to be reported in institutional units)

CONTACTS AND LOCATIONS:
Overall Officials: L E Hong, M.D., Principal Investigator — University of Maryland, Baltimore